CLINICAL TRIAL: NCT05158075
Title: Program for the Comprehensive Neurocognitive Treatment of Excess Weight
Acronym: TRAINEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raquel Vilar López (Other)
Collaborators: Ministerio de Ciencia, Innovación y Universidades, Spain (Unknown)
Responsible Party: Sponsor-Investigator, Raquel Vilar López, Principal Investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTI2018-098771-B-I00
Record Dates: First submitted 2021-11-17; First posted 2021-12-15 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Overweight
Keywords: Excess weight; Obesity; Overweight; Neurocognitive training
MeSH Terms: conditions — Obesity; Overweight | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The psychologists that conduct the assessments (screening, assessment sessions and follow-ups) will be blinded to the group allocation during the whole project. Moreover, since all assessments will be computerized and online, they are not subject to the biases of the evaluator. Further, all participants will be blind to their condition. Also, the people who perform the statistical analyses will be blind to the condition of the groups, through the coding of the interventions. Only the therapist performing the interventions will not be blind to the allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurocognitive training (Experimental): The experimental group will: i) receive three pre-treatment group sessions (Motivational Interviewing, nutrition and physical exercise); ii) receive an individualized diet and physical exercise planning for 6 weeks; iii) participate in 4 weekly group neurocognitive intervention sessions, that will last about 60-90 minutes each. Two neurocognitive sessions are intended to train impulsivity, and the other two neurocognitive sessions will focus on reflexive training. Participants will practice the content of each session daily at home.
  Interventions: Behavioral: Approach-Avoidance Bias Modification; Behavioral: Inhibition Training; Behavioral: Implementation of Intentions; Behavioral: Episodic Future Thinking; Behavioral: Motivational Interviewing; Behavioral: Nutritional intervention; Behavioral: Physical exercise intervention
- Sham cognitive training (Sham Comparator): The active control group will: i) receive three pre-treatment group sessions (Motivational Interviewing, nutrition and physical exercise); ii) receive an individualized diet and physical exercise planning for 6 weeks; iii) participate in 4 weekly group sessions of sham intervention that mimic the neurocognitive sessions of the experimental group. Two neurocognitive sessions are intended to train impulsivity, and the other two neurocognitive sessions will focus on reflexive training. Participants will practice the content of each session daily at home.
  Interventions: Behavioral: Sham Approach-Avoidance Bias Modification; Behavioral: Sham Inhibition Treatment; Behavioral: Setting Intentions; Behavioral: Recent Episodic Thinking; Behavioral: Motivational Interviewing; Behavioral: Nutritional intervention; Behavioral: Physical exercise intervention
- Control (Other): Participants in the control group will receive three pre-treatment group sessions (Motivational Interviewing, nutrition and physical exercise) and will receive an individualized diet and physical exercise planning for 6 weeks.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Nutritional intervention; Behavioral: Physical exercise intervention

INTERVENTIONS:
Behavioral: Approach-Avoidance Bias Modification — In this task participants must zoom in or zoom out a food image according to its format (vertical or horizontal) using their smartphone device. 90% of healthy food images will appear in the format to be approached (for example, vertical), while only 10% of unhealthy images will appear in that format (to ensure concentration on the task). The format to be approached will be counterbalanced. Participants will practice the task at home at least once a day (about 5 minutes) for one week, and will receive daily reminders to practice via instant messaging on their mobile phones.
  Other Names: Tilt Task
  Arms: Neurocognitive training
Behavioral: Inhibition Training — In this App participants are instructed to touch green circle items as quickly as possible, but to withhold their response and not to press on the red circle items, using their smartphone device. Some images are food, some non-foods. Participants can choose which food categories they would like to train to resist. The food-specific inhibition training condition included pictures of high-calorie foods always paired with the no-go signal. Participants will practice the task at least once a day (about 5 minutes) for one week, and will receive daily reminders to practice via instant messaging on their mobile phones.
  Other Names: Food Trainer
  Arms: Neurocognitive training
Behavioral: Implementation of Intentions — Participants establish one intention related to food and one related to exercise, and write when, where and how they will implement each one, possible inconveniences to do it, and how they will overcome them. Furthermore, motivational cues (why I eat) will be considered (negative emotions -I'm bored; social motives -eat a piece of cake you are offered in a party; politeness/conformity with others' expectations; pleasure). The implementation of intentions related to food will be written in format: "if… then…". This format allows for the consideration of the health goals and medium and long-term objectives for each of the participants. The intention related to food will focus on unhealthy snacking habits whenever possible. Participants will read and visualized their implementation of intentions at least twice a day (about 5 minutes) for one week, and will receive two daily reminders to practice via instant messaging on their mobile phones.
  Arms: Neurocognitive training
Behavioral: Episodic Future Thinking — Participants will decide health-related goals and anticipate positive future personal events at various time points (next month, 2-3 months and 4-6 months), from which contextual, temporal and emotional cues should be obtained. Goals and future events will be matched to generate episodic future thinking cues that include the necessary keys to facilitate their effectiveness. Participants will read and visualized their three cues at least twice a day (about 5 minutes) for one week, and will receive two daily reminders to practice via instant messaging on their mobile phones.
  Arms: Neurocognitive training
Behavioral: Sham Approach-Avoidance Bias Modification — Participants must zoom in or zoom out a food image according to the format (vertical or horizontal) using their smartphone device. 50% of healthy food images and 50% of unhealthy food images will appear in the format to be approached (for example, vertical). The format to be approached will be counterbalanced. Participants will practice the task at least once a day (about 5 minutes) for one week, and will receive daily reminders to practice via instant messaging on their mobile phones.
  Other Names: Sham Tilt Task
  Arms: Sham cognitive training
Behavioral: Sham Inhibition Treatment — In this App participants are instructed to touch green circle items as quickly as possible, but to withhold their response and not to press on the red circle items, using their smartphone devices. Some images are food, some non-foods. Participants can choose which food categories they would like to resist. High-calorie and low-calorie foods will be paired with the go signal on 50% of trials and with the no-go signal on 50% of trials. Participants will practice the task at least once a day (about 5 minutes) for one week, and will receive daily reminders to practice via instant messaging on their mobile phones.
  Other Names: Sham Food Trainer
  Arms: Sham cognitive training
Behavioral: Setting Intentions — Participants will choose 10 items of healthy foods to eat whenever they want to eat unhealthy food. They will also order a list of physical activities that they could do to lose weight. Participants will read their lists (food and exercise) at least twice a day (about 5 minutes) for one week, and will receive two daily reminders to practice via instant messaging on their mobile phones.
  Arms: Sham cognitive training
Behavioral: Recent Episodic Thinking — Participants will match habits and positive recent past events (1 day ago, 2 days ago, 1 week ago), both unrelated to food or physical activity, to establish their cues. Participants will read and visualized their three cues at least twice a day (about 5 minutes) for one week, and will receive two daily reminders to practice via instant messaging on their mobile phones.
  Arms: Sham cognitive training
Behavioral: Motivational Interviewing — Participants will assist a 90-minute group Motivational Interviewing session to maximize motivation and adherence to the program. The session will be guided through open questions and empathic reflections and affirmations to promote change talk. Participants will share their personal aims to reduce weight, improve their diet and increase their level of physical activity. Further, participants will talk about obstacles they have had on previous occasions, their expectations, and their motivations in regards to weight loss. When needed, information will be provided with the elicit-provide-elicit format. Sessions will end with an individual empathic summary for each participant's interventions.
Behavioral: Nutritional intervention — Participants will maintain a 60-minute group session with a nutritionist and will watch a 20-minute video to match and complete relevant information on nutrition. The nutritionist will design a 6-week individualized diet that participants will receive after the initial assessment. When the 6-week diet ends, participants will assist another 60-minute group session with the nutritionist and will watch another video intended to teach them how to design their own healthy diet and maintain long-term healthy eating habits.
Behavioral: Physical exercise intervention — Participants will maintain a 60-minute group session with a physical exercise professional and will watch a 20-minute video to match and complete relevant information on exercise. The physical exercise professional will design a 6-week physical exercise planning that participants will receive after the initial assessment. After those 6-weeks, participants will assist another 60-minute group session with the physical exercise professional and will watch another video intended to teach them how to design their own physical activity planning and maintain long-term healthy exercise habits.

SUMMARY:
The present study aims to determine the effectiveness of a comprehensive neurocognitive program for the treatment of excess weight. The program will include sessions to improve multiple cognitive processes implicated in weight gain and obesity. These cognitive processes include approach-avoidance bias, inhibition control, implementation intentions and episodic future thinking. Participants will be randomly allocated to one of three groups: 1) the experimental group will receive active neurocognitive sessions, 2) an active control group that will receive sham sessions and 3) a usual treatment control group. All three groups will receive a motivational interviewing session, along with personalized diet and physical exercise recommendations. We hypothesized that the neurocognitive program will decrease body mass index in people with overweight and obesity. In addition, the neurocognitive program will improve other anthropometric measures (waist circumference, waist-to-hip and waist-to-height ratios), lifestyle behaviors (eating behavior and physical activity), as well as cognitive processes (approach-avoidance bias, food inhibition, food liking and delay of gratification). Finally, the program will show its efficiency in the economic balance of cost-effectiveness and cost-utility.

DETAILED DESCRIPTION:
1. STARTING HYPOTHESES AND GENERAL OBJECTIVE HYPOTHESIS: The treatment of excess weight with a comprehensive program based on experimental knowledge about the functioning and modification of the impulsive and executive systems will be effective for the treatment of overweight and obesity. Thus, the neurocognitive training will reduce body mass index (BMI) in people with overweight and obesity, compared to a sham treatment and to only usual treatment. In addition, the neurocognitive program will improve other anthropometric measures (waist circumference, waist-to-hip and waist-to-height ratios), lifestyle behaviors (eating behavior and physical activity), as well as cognitive processes (approach-avoidance bias, food inhibition, food liking and delay of gratification). Finally, the program will show its efficiency in the economic balance of cost-effectiveness and cost-utility.

   GENERAL OBJECTIVE: To determine the effectiveness of a comprehensive neurocognitive program for the treatment of excess weight.

   1.1. Specific Aims: Objective 1: To examine the effectiveness of a comprehensive neurocognitive training to reduce BMI in the short, medium and long term (post-treatment, 3-month follow-up and 6-month follow-up).

   Objective 2: To study the effectiveness of the comprehensive neurocognitive program to change food behaviors, physical activity and body measures.

   Objective 3: To investigate which active ingredients have an impact on the results of the program as outlined below:

   3.1. To study the effectiveness of the impulsive training (approach-avoidance bias modification and improvement of inhibitory control) to reduce the approach bias to appetitive foods, increase the inhibitory control, improve the food decision making and modify the valuation of healthy and unhealthy foods.

   3.2. To study the effectiveness of reflexive training (implementation of intentions and episodic future thinking) to improve behaviors related to implementation of intentions in healthy eating and physical activity, and to increase delay of gratification.

   3.3. To compare the effectiveness of the neurocognitive training (impulsive and reflexive) to reduce BMI and body measures, and to improve food behaviors and physical activity.

   3.4. To study the variables related to cognition, affect, stress and non-homeostatic food intake, motivation and personality to predict or mediate the intervention results.

   Objective 4: To conduct an economic evaluation analysis of cost-effectiveness and cost-utility of the neurocognitive training in people with overweight and obesity, and analyze what budgetary impact would imply for the Spanish National Health System.
2. METHODOLOGY

   2.1. Design: Randomized controlled trial of parallel groups.

   2.2. Participants: The participants (N=150) will be randomly allocated to three groups: experimental group (neurocognitive intervention; n=50), active control group (sham intervention; n=50), and control group (treatment as usual; n=50).

   A randomization (minimization) through the software Minimizer® will be performed to avoid imbalances between the groups in age, sex, and BMI.

   2.3. Interventions: Pre-treatment interventions (all groups): Participants will participate in a group Motivational Interviewing session, and will receive an individualized diet and a physical exercise planning for 6 weeks. Also, informative videos and brochures will be provided. Further, participants will participate in two group informative sessions (one with a nutritionist and another with a physical exercise instructor). These two meetings will be recorded and made available for all participants.

   Whatsapp groups will be created to promote participants' social interactions.

   Neurocognitive program (experimental and active control groups). Duration: 4 weekly sessions of about 60-90 minutes.

   Phase 1. Impulsive training will include: (i) Approach-avoidance bias modification with the Tilt Task app; (ii) Inhibition training with the Food Trainer task app.

   Phase 2. Reflexive training will include: (iii) Implementation of Intentions; (iv) Episodic Future Thinking.

   The order of phases 1 & 2 will be counterbalanced. One task will be trained in each session, and participants will practice that task daily at home for one week (until the next session). They will receive daily reminders on their mobile phones. A weekly pre-post assessment will be conducted for each trained task.

   Post-treatment interventions (all groups): Participants will have the opportunity to attend a second group meeting with the nutritionist and another with the physical activity professional to receive information and ask questions about how to maintain long-term healthy habits on diet and physical exercise. These meetings will be recorded and made available for all participants. They will also be provided with new videos with guidelines about how to maintain a healthy long-lasting eating and exercise. The aim is that participants be autonomous and can develop their own diet and exercise planning.

   2.4. Outcome measures: Body Mass Index will be the main outcome measure. Secondary outcomes will measure changes in cognitive, lifestyle behaviors and body measures. Mediating and moderating variables will include affect, stress and nonhomeostatic eating, executive functions, motivation, personality, adherence to diet and physical exercise, and clinical variables. Further, assessment will include screening and descriptive variables, and measures to calculate cost-effectiveness, cost-utility and budget impact of the intervention program.
3. PROCEDURE All assessments and intervention sessions will be delivered online. Inclusion and exclusion criteria will be checked through the data collected in a questionnaire of sociodemographic and clinical variables. Further, psychopathology exclusion criteria will be tested with two questionnaires to measure depression, anxiety, and stress symptoms as well as binge eating and bulimia (DASS-21 and QEWP-5), and a short clinical interview by phone and/or information requested by email in those cases where there are doubts about any of the aspects collected through the online instruments.

All candidates who meet the criteria will attend an information meeting about the project in which they will receive written and oral information, and will be asked for their informed consent. Then, participants will be randomly assigned to groups before the pre-treatment assessment sessions. The three groups of the study (intervention, active control and control) will complete all of the evaluations, as well as the follow-ups (see below). Further, all groups will received the pre-treatment interventions (Motivational Interviewing, nutrition and physical activity sessions). What will differentiate the groups will be, therefore, the treatment: neurocognitive intervention vs. sham vs. usual treatment. The control groups will be offered the treatment sessions (without the assessment components) after the end of the 6-month follow-up.

Sessions will be developed in groups of 5-6 persons. If a participant misses a session he/she can attend another one within 3-4 days. There will be 10 experimental groups of active training = 50 participants; 10 active control groups of sham training = 50 participants; and 10 control groups = 50 participants. The program will comprise 8 weeks including three assessments (pre, intermedium and post-treatment), four intervention sessions, as well as pre-treatment and post-treatment intervention sessions. Also, two follow-up sessions at 3 and 6 months after treatment (see below). Sessions will last about 1 hour and a half.

Sessions will consist of the following:

1. Informative session (session 1; week 0): All participants will be informed about the aims and the procedure of the research, and they will provide written informed consent.
2. Pre-treatment assessment (session 2, week 1): All participants will complete the instruments to obtain the main and secondary outcomes, the potential mediators/moderators, and economic measures.
3. Pre-treatment interventions (sessions 3, 4 and 5, week 2):

   3.1. Motivational interviewing session: This 90-minute session will be developed in a group format of 5-6 participants.

   3.2. Nutrition session: Participants will receive an individualized diet for the following 6 weeks. Videos and brochures about nutrition will be provided, and participants will assist a 60-minute group session with the nutritionist to match and complete relevant information on nutrition and excess weight.

   3.3. Physical activity session: Participants will receive physical activity recommendations for the following 6 weeks. Videos and brochures about physical exercise will be provided, and participants will assist a 60-minute group session with the physical exercise instructor to match and complete relevant information on exercise and excess weight.
4. Intervention sessions (sessions 6, 7, 9 and 10; weeks 3, 4, 6 and 7): All sessions will start with Visual Analogue Scales to evaluate hunger, nutrition and physical activity. Each intervention session will be preceded by its pre-treatment evaluation, and followed by its post-treatment evaluation after a week of daily training. The pre and post-treatment evaluation of the impulsive training will be measured by the approach-avoidance bias (with the Tilt-Task app), food choice, the inhibitory control (with the Food Trainer app) and food liking. The pre and post-treatment evaluation of the reflexive training will be measured by the Now or Later questionnaire for the episodic future thinking training, and the self-registration of nutrition and physical exercise for the implementation of intentions.
5. Intermediate assessment (session 8; week 5): This assessment will allow the comparison between the interventions for the impulsive and reflexive trainings.
6. Post-treatment assessment (session 11, week 8): To evaluate the effectiveness of the whole intervention program, the measures of the pre-treatment assessment will be repeated.
7. Post-treatment interventions (session 12, week 8): After the post-treatment assessment, participants will have the opportunity to have a second 60-minute group meeting with the nutritionist and another with the physical activity professional, and they will be provided with new 20-minute videos about how to maintain a healthy long-lasting eating and exercise.

   After all interventions, participants will be asked to complete a debriefing to register their thoughts and subjective experience about the program.
8. Follow-up (sessions 13 and 14, week 20 and week 32): Follow-ups at 3 and 6 months after the intervention will include the instruments to obtain the main and secondary outcome measures. Besides, every month after the end of the treatment, participants will be contacted by email and mobile message to maintain adherence.

Participants will be instructed to eat two hours before all evaluation (pre, intermediate and post-treatment, and the two follow-ups) and neurocognitive sessions. Pre, intermediate and post-treatment assessments will be carried out at the same hour.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 39.9
* Age between 18 and 55 years
* Good command of the Spanish language
* Have at least two electronic devices available, one of them a smartphone with a gyroscope

Exclusion Criteria:

* Traumatic, digestive, metabolic or systemic disorders that affect the central nervous system, autonomic or endocrine
* Cardiovascular or any other disorders that prevent physical exercise
* Psychopathological disorders or presence of severe symptoms in the Depression Anxiety and Stress Scale-21 (DASS-21)
* Eating disorders or presence of criteria in the Questionnaire on Eating and Weight Patterns-5 (QEWP-5)
* Pharmacological or any other kind of treatment for losing weight at present
* Candidates for bariatric surgery
* Food conditions that could interfere with the stimulus of the program (allergies, spru, vegetarianism, veganism)
* Current pregnancy or breastfeeding (or expected pregnancy in the following six months)
* Weight loss >5% on the 3 months previous to the program
* Use of medication that affects weight
* Frequent use of alcohol or other drugs that affects food intake.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in Body Mass Index at post-intervention and follow-ups | Through study completion (8 months)
  Body mass index (BMI) is a measure of body fat based on height and weight. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m^2. Height and weight will be obtained with a pharmacy digital weight.

SECONDARY OUTCOMES:
Mean change from baseline in the Approach-avoidance bias on the Tilt Task app at 1 week | Counterbalanced week 3 or 6 (days 1 and 7)
  The Tilt Task average reaction time of the approach and avoidance trials will be subtracted separately for healthy and unhealthy foods, with the positive and negative scores representing approximation and avoidance bias, respectively. Reaction time will be measured before and after 1-week training.
Mean change from baseline in food inhibitory control on the Food Training app at 1 week | Counterbalanced week 4 or 7 (days 1 and 7)
  The Food Trainer app reaction time for the high-calorie and low-calorie foods paired with the go and the no-go signal will be measured before and after 1-week training. The average response time for go and no-go items will be calculated according to the type of images (appetizing and healthy foods), and commission errors will be recorded.
Mean change from baseline in food choice at post-intervention | Baseline (week 1), intermediate assessment (week 5) and post-treatment assessment (week 8)
  In the Food Choice task, 16 pictures of different healthy and unhealthy snack foods will be presented. Participants will select 8 of these foods. They will have 15 seconds to make their choices. The score will be the number of healthy foods selected.
Mean change from baseline in food liking at post-intervention | Baseline (week 1), intermediate assessment (week 5) and post-treatment assessment (week 8)
  Participants will be asked to imagine that different foods are in their mouth and to rate how much they like the taste with a visual analogue scale anchored at the extremes with "not at all" and "very much". Participants will move a cursor along the scale using a mouse and press the mouse button to confirm their rating, and the score between 0 and 100 will be recorded.
Mean change from baseline in delay of gratification on Now or Later at 1 week | Counterbalanced week 6 or 3 (days 1 and 7)
  Score on the questionnaire Now or Later will be used to measure the sensitivity relative to immediate rewards versus higher value rewards delayed at different time intervals. For the experimental group, each item of the questionnaire will be applied immediately after reading the episodic future thinking cue trained attending to the temporary interval of the item. For the active control group, each item of the questionnaire will be applied immediately after reading the recent episodic thinking cue trained attending to the temporary interval of the item. The control group will respond to the Now or Later questionnaire without any modification.
Mean change from baseline in Implementation of Intentions on a self-reported diary at 1 week | Baseline (week 1) and counterbalanced week 7 or 4 (days 1 to 7)
  Implementation of intentions will be assessed for 7 days with a self-reported diary to register frequency and quantity of foods in the snacking behavior, and frequency and time of physical exercise. The desire to snack and do physical exercise will be also recorded, as well as the achievement of intentions in the experimental/active control groups. For participants without snacking behaviors, personalized food goals will be used.
Mean change from baseline on a self-reported 72-hours intake foods at post-intervention and follow-ups | 8 months (at baseline-week 1-, weeks 5, 8, 20 and 32)
  Units and quantities on the amounts of foods and drinks that participants eat and drink during 72 hours will be transformed into total number of calories, as well as calories for carbohydrates, sugars and fat.
Mean change from baseline in healthy eating at post-intervention and follow-ups | Weeks 4, 5, 6, 7, 8, 20 and 32
  Participants will respond a Visual Analog Scale with the question: During the last week, how healthy do you think your diet has been? Healthy eating is understood as that according to the information received in the program: low amount of ultra-processed food, added sugar or alcohol; high amount of whole grain products, fruits and vegetables; etc. (0= no healthy at all; 100= 100% healthy).
Mean change from baseline in adherence to Mediterranean diet at post-intervention | Baseline (week 1) and post-treatment assessment (week 8)
  Mediterranean Diet Adherence Screener (MEDAS; Schröder et al., 2011): Score on the 14 items of the questionnaire that evaluate nutritional habits.
Mean change from baseline in the IPAQ at post-intervention and follow-ups | 8 months (at baseline-week 1-, weeks 5, 8, 20 and 32)
  International Questionnaire about physical activity (IPAQ; www.ipaq.ki.se): score on this questionnaire with 7 questions about physical activity during the last week, as well as time walking and sitting down.
Mean change from baseline in exercise habits at post-intervention and follow-ups | Weeks 4, 5, 6, 7, 8, 20 and 32
  Participants will respond a Visual Analog Scale with the question: During the last week, what has been your level of activity and physical exercise? (0= no activity at all; 100= maximum level of activity that I would be able to do).
Mean change from baseline in diary footsteps at post-intervention and follow-ups | Through study completion (8 months)
  A pedometer will be used to count diary steps
Mean change from baseline in waist circumference at post-intervention and follow-ups | 8 months (at baseline-week 1-, weeks 5, 8, 20 and 32)
  Participants should stand with heels close together and trunk erect, and put the tape measure around the waist, just above the navel, to measure the waist circumference in centimetres.
Mean change from baseline in waist-to-hip ratio at post-intervention and follow-ups | 8 months (at baseline-week 1-, weeks 5, 8, 20 and 32)
  Participants should stand with heels close together and trunk erect. To measure waist circumference, participants should put the tape measure around the waist, just above the navel. To measure hip circumference, participants should place the tape measure at the maximum gluteal prominence. The waist-to-hip ratio is determined by dividing the waist circumference (in cm) by the hip circumference (in cm).
Mean change from baseline in waist-to-height ratio at post-intervention and follow-ups | 8 months (at baseline-week 1-, weeks 5, 8, 20 and 32)
  Participants should stand with heels close together and trunk erect, and put the tape measure around the waist, just above the navel, to measure the waist circumference in centimeters. The height in centimeters will be measured with a digital weight. The waist to height ratio is determined by dividing the waist circumference by the height.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vilar-López, Ph.D., Principal Investigator — Universidad de Granada
Locations (1):
- Mind, Brain and Behavior Research Center at University of Granada (CIMCYC-UGR), Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee and who provide a methodologically sound proposal. Proposals should be directed to rvilar@ugr.es

REFERENCES:
- [Derived] Gonzalez-Gonzalez R, Solier-Lopez L, Vilar-Lopez R, Verdejo-Garcia A, Navarro-Perez CF, Caracuel A. Online Mental Contrasting with Implementation Intentions for changing snacking behavior and reducing body mass index in people with excess weight: a randomized controlled trial. Appetite. 2025 Oct 1;214:108209. doi: 10.1016/j.appet.2025.108209. Epub 2025 Jun 26. PMID 40581182
- See also: Web of the project — http://trainep.ugr.es/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT05158075/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT05158075/ICF_001.pdf